CLINICAL TRIAL: NCT06442189
Title: Prospective Evaluation of the Effects of the Mediterranean Diet on the Reproductive and Metabolic Parameters of Patients Diagnosed With Polycystic Ovary Syndrome (PCOS) and a Body Mass Indexof Over 25 kg/m2
Brief Title: The Results of the Mediterranean Diet for PCOS
Acronym: PCOS
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mujde Can Ibanoglu, Assoc. Prof, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: 01/06 22.01.2024
Record Dates: First submitted 2024-05-18; First posted 2024-06-04 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Polycystic Ovary Syndrome; Diet Habit
Keywords: polycystic ovary syndrome; Mediterranean diet; obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Feeding Behavior; Obesity | interventions — Diet, Mediterranean; BaseLine dental cement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3. month: Once the baseline values have been determined at the first visit, all tests are repeated after the diet has been followed for 3 months.
  Interventions: Dietary Supplement: Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: Mediterranean Diet — The aim was to evaluate the effects of the application of a Mediterranean diet on the reproductive and metabolic parameters in the 3rd month of patients with a body mass index of 25 and more who were treated in our clinic due to a diagnosis of PCOS.
  Other Names: Baseline; 3. Month

SUMMARY:
The aim was to evaluate the effects of the application of a Mediterranean diet on the reproductive and metabolic parameters in the 3rd month in patients with a body mass index of 25 and more who were followed up in our clinic due to a PCOS diagnosis.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is an endocrine-metabolic disorder characterized by menstrual irregularities, anovulation, clinical and/or biochemical symptoms of hyperandrogenism (hirsutism and/or acne), micropolycystic ovaries and metabolic abnormalities. Phenotype A: HA + OD + PCOM; phenotype B: HA + OD; phenotype C: HA + PCOM and phenotype D: OD + PCOM). According to the Rotterdam criteria, endocrine and metabolic abnormalities are lowest in the OD + PCOM group among these 4 different phenotype groups. The prevalence and distribution of metabolic abnormalities (insulin resistance, metabolic disease and glucose intolerance) among the phenotypes do not differ significantly between the 4 groups. Therefore, metabolic abnormalities and distribution characteristics are not suitable to distinguish different clinical PCOS phenotypes. Some inflammatory cytokines are elevated in PCOS, which is characterized by chronic low-grade inflammation. Although the exact mechanisms of inflammation in PCOS are not yet fully understood, it is thought to be mediated by obesity, insulin resistance and high androgen levels. This inflammatory state has a negative impact on the risk of future health problems and quality of life in PCOS. Therefore, strategies to reduce inflammation are considered important. Establishing medical nutrition therapy for PCOS has significant implications for reducing this inflammation and preventing the disease. At this point, the Mediterranean diet, which has been shown to have a protective effect against many diseases, is receiving a lot of attention. Among the components of the Mediterranean diet, omega-3 fatty acids, antioxidants and fiber in particular can contribute to reducing inflammation through various mechanisms. The international scientific community has strongly emphasized the role of the Mediterranean diet and the lifestyle it inspires in increasing life expectancy and improving public health. For these reasons, the Mediterranean diet can be considered as a nutrient pool containing nutraceuticals and bioactive components in foods that can positively influence health both directly and through their own epigenetic mechanisms. Recent studies suggest that the Mediterranean diet can influence both the incidence and severity of PCOS and the treatment of the disease.

The main objective of our study is to evaluate the effect of the MedDiet, which is known to be anti-inflammatory and based on energy restriction and the Mediterranean dietary approach, on the reproductive and metabolic parameters of PCOS patients with a higher than normal body mass index.

ELIGIBILITY:
Inclusion Criteria:

* At the age of 18-40 years,
* No underlying metabolic disease (type 2 diabetes, hypertension, diagnosed anemia),
* With a body mass index of 25 and above,
* Female patients attending the PCOS clinic and under the care of our hospital's dietitian will be enrolled in the study.

Exclusion Criteria:

1. Age < 18 and > 40 years;
2. Menopause, pregnancy or breastfeeding in the last 6 months;
3. Hyperandrogenism and/or biochemical hyperandrogenemia due to secondary etiologies, including congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome, hyperprolactinemia, thyroid dysfunction and adrenal disorders),
4. Pre-existing systemic or psychiatric disease
5. Use of drugs that affect carbohydrate or lipid metabolism (oral contraceptive pills, metformin, anti-epileptics, antipsychotics, statins and fish oil);
6. Certain eating regimens or hypocaloric diet in the last three months; supplementing with antioxidants, vitamins or minerals;
7. Non-steroidal anti-inflammatory drugs, diuretics, etc. use of medications that may affect fluid balance
8. Female patients with implanted pacemakers or defibrillators due to the theoretical possibility of interference with device activity.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People receiving care at the PCOS Clinic of Etlik Zübeyde Hanım Gynecology Training and Research Hospital who have a body mass index of 25 or more and follow a Mediterranean diet will be included in the study group.
  98 subjects who agreed to participate in the study and accepted the informed consent verbally and in writing will be included in the study. The study was designed to be prospective. Data will be collected after 0 and 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
the effect of applying a Mediterranean diet on Homa-IR in PCOS | 3 months
  Homeostasis model assessment (HoMA)-IR
PREDIMED in PCOS | 3 months
  PREDIMED questionnaire
the effect of applying a Mediterranean diet on glucose in PCOS | 3 months
  Fasting plasma glucose
the effect of applying a Mediterranean diet on HbA1c in PCOS | 3 months
  HbA1c values

CONTACTS AND LOCATIONS:
Overall Officials: Mujde Can Ibanoglu, Principal Investigator — Ankara Etlik Zubeyde Hanım Women's Health Training and Research Hospital, Ankara, Turkey.
Locations (1):
- Etlik Zübeyde Hanım, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Legro RS, Kunselman AR, Dodson WC, Dunaif A. Prevalence and predictors of risk for type 2 diabetes mellitus and impaired glucose tolerance in polycystic ovary syndrome: a prospective, controlled study in 254 affected women. J Clin Endocrinol Metab. 1999 Jan;84(1):165-9. doi: 10.1210/jcem.84.1.5393. PMID 9920077
- [Result] Barrea L, Arnone A, Annunziata G, Muscogiuri G, Laudisio D, Salzano C, Pugliese G, Colao A, Savastano S. Adherence to the Mediterranean Diet, Dietary Patterns and Body Composition in Women with Polycystic Ovary Syndrome (PCOS). Nutrients. 2019 Sep 23;11(10):2278. doi: 10.3390/nu11102278. PMID 31547562